CLINICAL TRIAL: NCT07338331
Title: Comparison Between the Effect of Aspirin and SGLT2 Inhibitor Intake in Non-Alcoholic Fatty Liver on Liver Enzymes, Lipid Profile, and the Results of FibroScan
Brief Title: Comparative Effects of Aspirin and SGLT2 Inhibitors on Liver Enzymes, Lipid Profile, and FibroScan Findings in Non-Alcoholic Fatty Liver Disease
Acronym: AS-NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galala University (Other)
Responsible Party: Principal Investigator, Eman Hamed, Lecturer of Clinical Pharmacy, Galala University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Galala U
Record Dates: First submitted 2025-12-20; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Diabete Type 2; Non Alcoholic Fatty Liver
Keywords: Non-alcoholic fatty liver disease, Aspirin, Dapagliflozin, Liver enzymes, Lipid profile
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — Aspirin; dapagliflozin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aspirin group (Experimental): Participants were received 100 mg of aspirin as oral daily doses for 6 months.
  Interventions: Drug: Aspirin
- Dapagliflozin group (Experimental): Participants were received 10 mg of dapagliflozin as oral once-daily doses for 6 months.
  Interventions: Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy

INTERVENTIONS:
Drug: Aspirin — Participants received 100 mg of aspirin (aspirin protect®) as oral daily doses for 6 months.
  Other Names: aspirin protect®
  Arms: aspirin group
Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy — Participants received 10 mg of dapagliflozin (Diaflozimet ®) as oral once-daily doses for 6 months.
  Other Names: Diaflozimet ®
  Arms: Dapagliflozin group

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a prevalent hepatic manifestation of metabolic syndrome, encompassing a spectrum of liver disorders from steatosis to non-alcoholic steatohepatitis (NASH), with potential progression to advanced fibrosis, cirrhosis, and hepatocellular carcinoma. Given the global health burden of NAFLD, therapeutic interventions targeting its pathophysiological mechanisms are crucial.

DETAILED DESCRIPTION:
A randomized, controlled clinical trial will be conducted over 6 months with 80 participants diagnosed with NAFLD. Participants will be assigned to one of the groups including the Aspirin group (100 mg/day), and Empagliflozin 10 mg once daily. Primary outcomes include changes in liver enzymes, lipid profiles, and Fibroscan results, while secondary outcomes focus on clinical symptoms and metabolic indicators like body weight and waist circumference.

Statistical Analysis: Paired t-tests will compare pre- and post-treatment values within each group, while independent t-tests will assess differences between groups. A significance level of p<0.05 will be used.

ELIGIBILITY:
Inclusion Criteria: if one or more the following are present:

* Diabetes mellitus, unless receiving only Dapagliflozin for treatment.
* Adult individuals (18-65 years) with a clinical diagnosis of NAFLD based on liver ultrasound
* No history of alcohol consumption or consumption within 3 months.
* Absence of other liver diseases.
* No significant renal or gastrointestinal issues that could interfere with treatment.

Exclusion Criteria:Patients were excluded from our study if one or more the -following are present:

* Pregnancy or breastfeeding.
* Active chronic viral hepatitis or autoimmune liver disease.
* History of gastrointestinal bleeding or other contraindications for Aspirin.
* Severe renal insufficiency.
* Alcohol intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
lipid profile and Fibroscan results | 6 months
  * Changes in liver enzymes (AST, ALT, ALP, GGT) after 6 months.
  * Lipid profile (Total Cholesterol, LDL, HDL, Triglycerides) at baseline and after 6 months.
  * Fibroscan results (liver stiffness measurement) at baseline and after 6 months.
lipid profile and Fibroscan evalution | 6 months
  * Changes in liver enzymes (AST, ALT, ALP, GGT) after 6 months.
  * Lipid profile (Total Cholesterol, LDL, HDL, Triglycerides) at baseline and after 6 months.
  * Fibroscan results (liver stiffness measurement) at baseline and after 6 months.

SECONDARY OUTCOMES:
indicators of metabolic improvement | 6 months
  * Improvement in clinical symptoms (fatigue, discomfort).
  * Impact on body weight and waist circumference (as indicators of metabolic improvement).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No